CLINICAL TRIAL: NCT01766232
Title: Lacrimal Drainage Resistance Study
Acronym: LDRS
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Julian Perry, MD, The Cleveland Clinic
Other Study IDs: IRB 07-926
Record Dates: First submitted 2011-05-13; First posted 2013-01-11 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Epiphora; Nasolacrimal Duct Obstruction; Canalicular Stenosis; Functional Tear Pump Failure; Ectropion
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Lacrimal Duct Obstruction; Ectropion

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obstructed nasolacrimal drainage group: This group of patients is clinically identified as having epiphora due to an obstruction of the lacrimal drainage system.
- Ectropion group: This group of patients is clinically determined to have functional epiphora due to ectropion and a patent lacrimal drainage system.

SUMMARY:
Epiphora, or uncontrolled tearing of the eyes, represents a common presenting complaint of patients seen by ophthalmologists. Epiphora may be due to non-obstructive causes, such as tear hypersecretion or functional tear pump failure, or obstructive causes. Functional tear pump failure may result from malposition of the eyelids, such as an abnormal out-turning (ectropion) or in-turning (entropion) of the eyelid.

Currently methods to diagnose partial nasolacrimal duct obstruction are purely qualitative in nature. Our research goal is to quantitatively measure the pressure generated during conventional probing and irrigation (P&I), and to measure the resistance to irrigation of the nasolacrimal drainage system.

The investigators will measure the pressure generated during conventional P&I using a disposable in-line pressure transducer. In addition, the investigators will use a syringe pump to deliver a constant flow rate of saline through a nasolacrimal cannula and measure the steady state irrigation pressure using the in-line transducer and digital pressure monitor. Resistance can be directly calculated from the known flow rate and pressure measurements.

The investigators will compare both the pressure generated during P&I and the lacrimal drainage resistance between patients with lacrimal drainage obstruction and controls patients with no obstruction (functional tear pump failure) as determined by clinical exam.

Clinical applications for measuring lacrimal drainage resistance include quantifying partial nasolacrimal duct obstruction, guiding the choice of surgical procedure, and determining the success of lacrimal drainage procedures.

DETAILED DESCRIPTION:
Lacrimal Drainage Resistance

I. Introduction

This proposal describes our plan to study the resistance of the lacrimal drainage system during irrigation.

II. Research Aims

A. Specific Aims

1. To quantitatively measure the resistance of the lacrimal drainage system during irrigation.
2. To determine differences in lacrimal drainage resistance between patients with obstructed tear drainage systems and patients with functional tear pump failure.
3. To measure the pressure generated during traditional probing and irrigation of the lacrimal drainage system.

B. Background and Significance

Epiphora, or uncontrolled tearing of the eyes, represents a common presenting complaint of patients seen by ophthalmologists. Epiphora may be due to non-obstructive causes, such as tear hypersecretion or functional tear pump failure, or obstructive causes. Functional tear pump failure may result from malposition of the eyelids, such as an abnormal out-turning (ectropion) or in-turning (entropion) of the eyelid.

Tears normally drain from the eye through two small holes, called puncta, one located in the upper eyelid and one in the lower eyelid, and then through two channels, called canaliculi, that empty into the lacrimal sac. Tears drain from the lacrimal sac through the bony nasolacrimal duct into the nasal cavity. Obstruction may occur at any level of the system, and may be partial or complete.[1] The focus of this study is acquired (as opposed to congenital), nasolacrimal duct obstruction.

The normal work-up for evaluation of nasolacrimal duct obstruction includes multiple clinical tests to evaluate the patency of the drainage system, including the fluorescein dye disappearance test, primary and secondary Jones dye tests, and canalicular probing and irrigation (P&I). While complete obstruction is relatively easily determined, partial obstruction is more difficult. Each of the available tests is qualitative in nature and is unable to determine the degree of partial obstruction. [1, 2] Current management options for the treatment of partial nasolacrimal duct obstruction include repeated canalicular probing and irrigation, balloon catheter dilation with placement of silicone stents, and dacryocystorhinostomy (DCR) surgery. Repeated probing and irrigation may be performed in the clinic without anesthesia, but has a low rate of improved symptoms. Balloon catheter dilation with stent placement is typically performed under general anesthesia, requires no incisions, and has a success rate between 60-73%.[3, 4]. DCR surgery, also typically performed under general anesthesia, surgically bypasses the nasolacrimal duct by removing a window of bone and anastomosing the lacrimal sac to the nasal cavity. The success rate of DCR is over 95%.[1, 5] There are two previously published methods to measure lacrimal drainage resistance. In 1991, Stanley and Masri described a device to measure resistance with a hand-held instrument connected to a personal computer.[6] They reported values from 13 normal controls, but did not test the device in patients with tearing. In 1995, Tucker et al. reported a laboratory-based device that measured the resistance to fluid flow in the lacrimal drainage system.[2] They measured resistance in healthy controls, in patients after successful DCR, and in one tearing patient.

The investigators will measure the pressure generated during conventional P&I using a disposable in-line pressure transducer. In addition, the investigators will use a syringe pump to deliver a constant flow rate of saline through a nasolacrimal cannula and measure the steady state irrigation pressure using the in-line transducer and digital pressure monitor. Resistance can be directly calculated from the known flow rate and pressure measurements.

Clinical applications for measuring lacrimal drainage resistance include quantifying partial nasolacrimal duct obstruction, guiding the choice of surgical procedure, and determining the success of lacrimal drainage procedures.

III. Study Design and Methods

Study Design:

The investigators plan to measure lacrimal drainage resistance in consented patients undergoing evaluation and management of epiphora who require traditional probing and irrigation. In addition to the traditional probing and irrigation of the nasolacrimal system, the investigators will measure the lacrimal drainage resistance using our study equipment.

Accrual Goals and Recruitment Period:

The accrual goal for this study is 40 eligible patients.

The final clinical diagnosis of lacrimal drainage obstruction versus functional tear pump failure will be based upon the investigators clinical findings and standard probing and irrigation results.

Patient Entry:

Patient eligibility will be determined by the study's principal investigator or co-investigators and as described in this protocol. The investigator will interview eligible patients and explain in detail the purpose of the study. Those patients who agree to participate will have the pressure measured during conventional P&I and lacrimal drainage resistance measured in addition to the normal clinical work-up. For those patients who agree to participate in the study, signing the informed consent constitutes study entry.

Time Requirement:

The investigators estimate that it will take 2 months for patient accrual and measurements.

Follow-Up:

There are no required follow-up visits.

Measurement of outcomes:

Two measurements will be obtained from each patient. First, the investigators will record the pressure generated during traditional probing and irrigation using a disposable in-line pressure transducer. Second, the investigators will measure the pressure generated using a syringe pump to deliver a constant flow rate. The investigators will then directly calculate the resistance to irrigation from the pressure and flow rate.

IV. Study Procedure: The Intervention

Probing and irrigation (P&I) of the lacrimal drainage system is a standard component of the evaluation of tearing patients. During this procedure, a nasolacrimal cannula is inserted into the canaliculus and saline solution is irrigated through the system. The investigators will measure the pressure generated during P&I using a disposable in-line pressure transducer. In addition to conventional P&I, consented patients would undergo a second irrigation procedure using our measuring equipment. In order to eliminate any bias due to the order of testing, half of the patients will undergo conventional P&I first, and half will undergo the experimental P&I first. During the experimental P&I, a syringe pump will deliver a constant flow rate of saline through a nasolacrimal cannula. The investigators will measure the steady state irrigation pressure using an in-line transducer and digital pressure monitor. Resistance will be calculated from the known flow rate and pressure measurements. The investigators will obtain three measurements from each patient.

The syringe pump is designed to prevent backflow of saline, and in addition the disposable portion of the pressure transducer exposed to the saline will be changed between each patient. The syringe pump has an automatic safety cut-off if the line is occluded.

V. Interpretation of Data

The investigators will record the pressure generated during conventional P&I and the average pressure generated during steady-state irrigation. Resistance will be directly calculated from the average pressure measurement. The investigators will compare both the pressure generated during P&I and the lacrimal drainage resistance between patients with lacrimal drainage obstruction and controls patients with no obstruction (functional tear pump failure) as determined by clinical exam. The investigators will summarize data in terms of means and standard deviations. The null hypothesis, that there are no differences between groups, will be tested by a two-sample Students t-test with p < .05 for rejection of the null. For lacrimal drainage resistance, a sample size of 17 patients per group gives a power of 0.91 to detect a difference as small as 20 mmHg*sec/ml. The power measurements are based upon the work of Tucker et al., who measured an average resistance of 49.5 +/- 17.0 mmHg*sec/ml in normal controls, and a single measurement of 212 mmHg*sec/ml in a patient with symptomatic tearing.[2] Technical complications will be noted and described. All patient information will be a part of the permanent medical record and will be no different from the information documented in standard nasolacrimal irrigation.

VI. Consent Procedure

In addition to a verbal discussion describing the study, including the risks and benefits, the investigators will provide patients undergoing evaluation for epiphora including conventional probing and irrigation with a formal consent form, and the investigators will provide a copy of this consent for personal reference. The proposed consent form is attached.

VII. Adverse Events

The anticipated adverse events of conventional probing and irrigation are anxiety and discomfort during the procedure, foreign body sensation for 12-24 hours following the procedure, and irrigant or dye on clothing. Anticipated serious adverse events of conventional probing and irrigation include dacryocystitis and damage to the lacrimal drainage system including punctal rupture. The incremental risks of the experimental probing and irrigation relate to the pump device. Because the pump device has an automatic safety cut-off and pushes fluid at a very low flow rate (0.09 mL/s) the investigators believe that the incremental risks are very low. Stanley and Masri reported one case of punctal rupture using their experimental setup.[6] The investigators believe this is unlikely to occur in our experiment because the investigators are using a standard nasolacrimal cannula to irrigate, and the investigators are using a much lower flow rate (0.09 mL/s versus 0.25 mL/s).

All adverse events will be documented in the data collection forms and brought to the attention of the patient and his or her family as soon as possible after their occurrence. Patients are provided with contact information for the principle investigator as well as the Institutional Review Board in the consent form, and an on-call ophthalmologist is always available for emergent care after hours. On-call ophthalmologists will have direct pager access to the investigators and will notify them immediately of any adverse events encountered in study patients. Serious and unanticipated adverse events will be promptly reported to the Institutional Review Board by the principle investigator.

VII. Cited Literature

1. Mills, D.M. and D.R. Meyer, Acquired nasolacrimal duct obstruction. Otolaryngol Clin North Am, 2006. 39(5): p. 979-99, vii.
2. Tucker, S.M., et al., Measurement of the resistance to fluid flow within the lacrimal outflow system. Ophthalmology, 1995. 102(11): p. 1639-45.
3. Kuchar, A. and F.J. Steinkogler, Antegrade balloon dilatation of nasolacrimal duct obstruction in adults. Br J Ophthalmol, 2001. 85(2): p. 200-4.
4. Perry, J.D., et al., Balloon catheter dilation for treatment of adults with partial nasolacrimal duct obstruction: a preliminary report. Am J Ophthalmol, 1998. 126(6): p. 811-6.
5. Tsirbas, A., G. Davis, and P.J. Wormald, Mechanical endonasal dacryocystorhinostomy versus external dacryocystorhinostomy. Ophthal Plast Reconstr Surg, 2004. 20(1): p. 50-6.
6. Stanley, C.F. and F.A. Masri, Instrument to test patency of lacrimal drainage system. J Clin Eng, 1991. 16(1): p. 57-60.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) who present for evaluation of epiphora due to obstructed causes, and control patients who present for evaluation of epiphora due to non-obstructed functional causes, who have been recommended for traditional probing and irrigation

Exclusion Criteria:

* Active infection
* Punctal stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the oculoplastics service with epiphora.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lacrimal drainage resistance | one-time clinical measurement

SECONDARY OUTCOMES:
Pressure generated during nasolacrimal duct irrigation | one-time clinical measurement

CONTACTS AND LOCATIONS:
Overall Officials: Julian D Perry, MD, Principal Investigator — Cleveland Clinic Cole Eye Institute; Brian Costin, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Cole Eye Institute, Cleveland, Ohio, United States

REFERENCES:
- [Background] Kuchar A, Steinkogler FJ. Antegrade balloon dilatation of nasolacrimal duct obstruction in adults. Br J Ophthalmol. 2001 Feb;85(2):200-4. doi: 10.1136/bjo.85.2.200. PMID 11159486
- [Background] Mills DM, Meyer DR. Acquired nasolacrimal duct obstruction. Otolaryngol Clin North Am. 2006 Oct;39(5):979-99, vii. doi: 10.1016/j.otc.2006.07.002. PMID 16982258
- [Background] Perry JD, Maus M, Nowinski TS, Penne RB. Balloon catheter dilation for treatment of adults with partial nasolacrimal duct obstruction: a preliminary report. Am J Ophthalmol. 1998 Dec;126(6):811-6. doi: 10.1016/s0002-9394(98)00278-5. PMID 9860005
- [Background] Stanley CF, Masri FA. Instrument to test patency of lacrimal drainage system. J Clin Eng. 1991 Jan-Feb;16(1):57-60. doi: 10.1097/00004669-199101000-00014. PMID 10109831
- [Background] Tsirbas A, Davis G, Wormald PJ. Mechanical endonasal dacryocystorhinostomy versus external dacryocystorhinostomy. Ophthalmic Plast Reconstr Surg. 2004 Jan;20(1):50-6. doi: 10.1097/01.IOP.0000103006.49679.23. PMID 14752311
- [Background] Tucker SM, Linberg JV, Nguyen LL, Viti AJ, Tucker WJ. Measurement of the resistance to fluid flow within the lacrimal outflow system. Ophthalmology. 1995 Nov;102(11):1639-45. doi: 10.1016/s0161-6420(95)30815-9. PMID 9098256